CLINICAL TRIAL: NCT05247463
Title: Observational Study of Age, Test THreshold and Frequency on English NAtional Mammography Screening Outcomes (ATHENA-M)
Brief Title: English Mammography Screening Outcomes by Age, Frequency and Test Threshold
Acronym: ATHENA-M
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Warwick (Other)
Collaborators: University of Birmingham (Other); University of Bristol (Other)
Responsible Party: Principal Investigator, Sian Taylor-Phillips, Professor of Population Health, University of Warwick
Other Study IDs: SOC.03/20-21
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Screening; Observational
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women invited to Breast Cancer Screening in England: Women invited to Breast Cancer Screening in England up to 31st March 2018
  Interventions: Other: Increase in upper age of eligibility for breast cancer screening from 64 to 70
- Women attending Breast Cancer Screening in England: Women attending mammography screening to examine the effect of screening test threshold on outcomes, up to 31st March 2018
  Interventions: Other: Screening round length; Diagnostic Test: Screening test threshold

INTERVENTIONS:
Other: Increase in upper age of eligibility for breast cancer screening from 64 to 70 — The upper age limit of eligibility for Breast Cancer Screening increased in England from 64 to 70 as a result of the NHS Cancer Plan, so women were offered an additional 2 rounds of screening.
  Groups: Women invited to Breast Cancer Screening in England
Other: Screening round length — The target round length (frequency) of breast cancer screening in England is every 3 years. However in practice there is variability in this due to local centre capacity. The exposures are round lengths of approximately 2 years and approximately 3 years
  Groups: Women attending Breast Cancer Screening in England
Diagnostic Test: Screening test threshold — Radiologists and equivalent health professionals examine women's screening mammograms for potential signs of cancer, and recall some women for further diagnostic tests. Each has a different test threshold for recall, characterised by the proportion of previous cases that they have recalled.
  Groups: Women attending Breast Cancer Screening in England

SUMMARY:
Breast cancer screening involves taking mammograms (x-rays) of women's breasts to search for signs of cancer. This study investigates the impact of test threshold, screening interval (frequency) and age of eligibility on intermediate outcomes, and health outcomes such as mortality and morbidity. This observational study links breast cancer screening, cancer registry and mortality registration data to answer these questions.

DETAILED DESCRIPTION:
Breast cancer screening involves taking mammograms (x-rays) of women's breasts to search for signs of cancer. Different countries give different versions of breast screening, because there is no clear evidence which is best. This study investigates the effect of three variations to breast screening on outcomes for women screened.

Firstly, the test threshold. When radiologists examine the women's mammograms it is often not clear whether cancer is present. The test threshold means the tendency of radiologists to recall more or fewer women for further tests. In England overall 4% of women are recalled for further tests because their mammograms show suspicious signs, but different radiologists vary between 2% and 10%. This study investigates how recalling different proportions of women affects their long term outcomes.

Secondly the interval between screening invitations. In the UK breast screening is every 3 years, which is the longest time between screens in the world. In the US it is every year or 2 years and in Europe every 2 years. This study uses the natural variation in English screening interval to investigate the impact on women's outcomes.

Thirdly the age women are invited for breast screening. The NHS Cancer Plan in England resulted in extension of the upper age limit of eligibility for breast cancer screening from 64 to 70. This study investigates the change on women's outcomes.

The primary outcomes are health outcomes or close approximations, such as mortality, overdiagnosis of cancer which would never have caused harm, stage shift in cancer diagnosis, treatment (to reflect treatment associated morbidity), and false positive recall to assessment (which is known to induce anxiety). Secondary outcomes are intermediate outcomes with known but more proximal links to health outcomes: number of cancers detected at screening and their characteristics, and number of interval cancers detected between screening rounds.

This is an observational study linking women's screening records to cancer registry and mortality records from 1988 to 2018.

This observational study began on 1st January 2021, building on the POSTBOx study (NCT04365114). POSTBOx evaluates the impact of one or two readers on women's outcomes, POSTBOx primary outcomes 4 and 5 and secondary outcome 1 were dependent on obtaining follow up funding, which was achieved in this ATHENA-M project. The ATHENA-M funding also adds two additional exposures (screening interval and age of eligibility), and expands analysis of the test threshold exposure. Both projects were significantly delayed in data linkage and transfer, the investigators expect complete data transfer to the analysis team at Warwick between February and April 2022.

ELIGIBILITY:
Inclusion Criteria:

* Women invited for breast cancer screening by the English NHS Breast Screening Programme

Exclusion Criteria:

* Missing or corrupted data for NHS number, so linkage between databases is not possible
* For analysis of test threshold and screening interval: women who did not attend routine English NHS Breast screening service within the specified date and age range, even if they attended symptomatic breast cancer services, high risk (family history) breast screening services, or if they were referred for mammograms by their general practitioner

Ages: 47 Years to 73 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women invited for a Breast Cancer Screening appointment in England between 1st January 1988 and 31st March 2018. For test threshold and screening interval data this is further limited to women attending at least one breast screening appointment meeting the age and date eligibility requirements. The population will be further limited to women invited for breast cancer screening after 1st January 1998, if accurate data linkage cannot be achieved before this date in the absence of a unique identifier (before the widespread implementation of NHS number)
Sampling Method: Probability Sample
Enrollment: 10000000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Breast Cancer Specific Mortality | Cumulative incidence of breast cancer specific mortality over all follow-up time (up to maximum 30 years)
  Breast Cancer Specific Mortality
Breast Cancer Specific Mortality | 10 year follow up of particular importance to match previous systematic review of results
  Breast Cancer Specific Mortality
Breast Cancer Specific Mortality | 13 year follow up of particular importance to match previous systematic review of results
  Breast Cancer Specific Mortality
All cause mortality | Cumulative incidence of all-cause mortality over all follow-up time (up to maximum 30 years)
  All cause mortality
All cause mortality | 10 year follow up of particular importance to match breast cancer mortality
  All cause mortality
All cause mortality | 13 year follow up of particular importance to match breast cancer mortality
  All cause mortality
Overdiagnosis | Cumulative incidence of cancer over all follow-up time (up to maximum 30 years)
  Overdiagnosis of breast cancer which would not have been detected symptomatically using compensatory drop method, (difference between cumulative incidence of cancer (screening and symptomatic) between exposure groups
Overdiagnosis | 10 year follow up of particular importance to match breast cancer mortality
  Overdiagnosis of breast cancer which would not have been detected symptomatically using compensatory drop method, (difference between cumulative incidence of cancer (screening and symptomatic) between exposure groups
Overdiagnosis | 13 year follow up of particular importance to match breast cancer mortality
  Overdiagnosis of breast cancer which would not have been detected symptomatically using compensatory drop method, (difference between cumulative incidence of cancer (screening and symptomatic) between exposure groups
Stage Shift | For breast cancers detected at any point during follow-up (up to a maximum 30 years)
  Difference in prognostic indicators (DCIS vs invasive, grade, size, nodes involved, cancer type, hormonal status, Nottingham Prognostic Index, distant metastasis) between exposure groups, including both symptomatically and screen detected cancers
Treatment Received | Within 1 year of diagnosis
  Breast Cancer Treatment received (as a proxy for treatment associated morbidity)
False positive recall to assessment | At point of screening episode
  Proportion of women recalled for further tests from their screening mammogram, in whom those further tests did not detect breast cancer

SECONDARY OUTCOMES:
Interval cancers | Up to 3 years after the screening appointment
  Biopsy-proven breast cancers detected after symptomatic referral during the time interval between screening mammograms.
Cancers detected at screening | At screening episode
  Number of biopsy proven cancers detected at screening (• Definition includes any invasive cancer or Ductal Carcinoma in situ (DCIS) or Lobular Carcinoma in Situ (LCIS) of the breast, using standard definition of cancer registry and screening programme) with subgroup with invasive cancer only also reported
Screen detected cancer characteristics | At screening episode
  (DCIS vs invasive, grade, size, nodes involved, cancer type, hormonal status, Nottingham Prognostic Index, distant metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Warwick, Coventry, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The investigators do not have Office for Data Release permissions to share these data more widely, but can assist other researchers in applying for access.

DOCUMENTS (1):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT05247463/Prot_000.pdf